CLINICAL TRIAL: NCT06485245
Title: A Phase I Study Evaluating the Safety, Tolerability, Pharmacokinetics and Food Effect of Randomized, Double-Blind, Placebo-Controlled Single and Multiple Dose Escalations of CS060304 in Healthy and Elevated LDL-C Subjects
Brief Title: Study to Evaluate Safety, Tolerability and Pharmacokinetics of CS060304 in Healthy and Elevated LDL-C Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cascade Pharmaceuticals, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS060304-FIH-CN-I-01
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: MASH

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Cohort A1: 0.2mg CS060304 (Experimental): Healthy subjects in a fasting state will receive a single dose of CS060304 0.2 mg or placebo.
  Interventions: Drug: CS060304
- Cohort A2: 1mg CS060304 (Experimental): Healthy subjects in a fasting state will receive a single dose of CS060304 1 mg or placebo.
  Interventions: Drug: CS060304
- Cohort A3: 4mg CS060304 (Experimental): Healthy subject in fasted state receive a single oral dose of CS060304 4 mg or placebo on day 1, followed by a 4 day washout period, subjects in fed state will receive the same single oral dose of CS060304 4mg or placebo on day 5.
  Interventions: Drug: CS060304
- Cohort A4: 10mg CS060304 (Experimental): Healthy subjects in a fasting state will receive a single dose of CS060304 10 mg or placebo.
  Interventions: Drug: CS060304
- Cohort A5: 20mg CS060304 (Experimental): Healthy subjects in a fasting state will receive a single dose of CS060304 20 mg or placebo.
  Interventions: Drug: CS060304
- Cohort A6: 40mg CS060304 (Experimental): Healthy subjects in a fasting state will receive a single dose of CS060304 40 mg or placebo.
  Interventions: Drug: CS060304
- Cohort B1: 2mg CS060304 (Experimental): Elevated LDL-C subjects will receive the CS060304 2 mg or placebo once daily for a consecutive 14 days.
  Interventions: Drug: CS060304
- Cohort B2: 5mg CS060304 (Experimental): Elevated LDL-C subjects will receive the CS060304 5 mg or placebo once daily for a consecutive 14 days.
  Interventions: Drug: CS060304
- Cohort B3: 10mg CS060304 (Experimental): Elevated LDL-C subjects will receive the CS060304 10 mg or placebo once daily for a consecutive 14 days.
  Interventions: Drug: CS060304
- Cohort B4: 20mg CS060304 (Experimental): Elevated LDL-C subjects will receive the CS060304 20 mg or placebo once daily for a consecutive 14 days.
  Interventions: Drug: CS060304

INTERVENTIONS:
Drug: CS060304 — Tablets administered orally
  Other Names: Pleacbo

SUMMARY:
Study to Evaluate Safety, Tolerability and Pharmacokinetics of CS060304 in Healthy and Elevated LDL-C Subjects.

DETAILED DESCRIPTION:
A Phase I study Evaluating the Safety, Tolerability, Pharmacokinetics and Food Effects of Randomised, Double-Blind, Placebo-Controlled Single and Multiple Dose Escalations of CS060304 in Healthy and Elevated LDL-C Subjects.

ELIGIBILITY:
Inclusion Criteria:

SAD

1. Sign and date the ICF.
2. Signing ICF age≥18 years≤55 years, male or female.
3. Weight: Male≥50kg, female≥45kg BMI: 18~28kg/m².
4. Female or male subjects must be eligible for contraception during the study and for three months after the last dose.
5. Normal renal function.
6. Good general health.
7. No significant medical history, in good general health as assessed by the study during the Screening Period and no more than 28 days from the first dose.
8. Understand and comply with study procedures and limitations.

MAD

1. Sign and date the ICF.
2. Signing ICF age≥18 years≤65 years, male or female.
3. Weight: Male≥50kg, female≥45kg BMI: 18~35kg/m².
4. Screening period, fasting LDL-C > 110 mg/dL (2.85 mmol/L).
5. Female or male subjects must be eligible for contraception during the study and for three months after the last dose.
6. Normal renal function.
7. Good general health.
8. No significant medical history, in good general health as assessed by the study during the Screening Period and no more than 28 days from the first dose.
9. Understand and comply with study procedures and limitations. -

Exclusion Criteria:

SAD

1. Special dietary requirements, not following a uniform diet.
2. Pregnant or nursing females or females who have pregnancy plans during the trial or within 3 months after the trial.
3. History of febrile illness or active infection within 7 days prior to first dose.
4. Positive urine drug screens at screening or baseline.
5. History of substance/drug abuse in the 5 years prior to the start of the trial, or a positive screening or baseline drug screen result.
6. History of previous corrected QT interval (QTc) prolongation:

   1. Screening periods QTcF ≥ 450 ms.
   2. Family history of hypocalcaemia or long QT interval syndrome.
   3. Use of drugs causing QT/QTc prolongation.
   4. Investigator judgement of clinically significant abnormal ECG results.
7. Abnormal liver function: AST, ALT, ALP, GGT and TBIL>ULN.
8. Smoking or use of nicotine products within 3 months prior to screening and during the study period.
9. Use of other investigational drugs 40 days prior to enrolment or within at least 5 half-lives of drug use.
10. Positive screening results for infectious diseases during the screening period, include HIV, HBsAg, HBcAb, HCV antibody tests.
11. Any abnormal results of laboratory tests judged by the investigator to be clinically significant during the screening period.
12. Blood loss within 40 days prior to administration 50~500 mL, or loss of more than 500 mL of blood within 56 days prior to administration.
13. Men and women who consumed more than 1 unit per day prior to screening. [1 unit = 150 ml of wine, 360 ml of beer or 45 ml of 40% alcohol]. Subjects will not be permitted to consume alcohol 48 hours prior to dosing and while in the CRU.
14. Prescription and over-the-counter use within 14 days or at least 5 half-lives prior to the baseline period, or use of any drug or other substance that may affect CYP3A activity within 14 days or at least 5 half-lives before taking this study drug.
15. History of thyroid disease or clinically significant thyroid test abnormalities.
16. Allergy to thyroid medication.
17. Presence of any disease that may interfere with the absorption, distribution, metabolism or excretion of drugs, Including bile salt metabolism in the colon, such as gastrectomy, inflammatory bowel disease, etc.
18. According to the researcher's judgment, there are clinically significant diseases found, including but not limited to (gastrointestinal, kidney, liver, nervous, blood, endocrine, tumor, lung, immune, mental or cardiovascular diseases), researchers believe that participating in the study poses risks to participants.
19. Allergy to the investigational drug or any component of the investigational drug, Allergy history and constitution.
20. Diseases or conditions with clinical significance that researchers believe may pose a risk to the safety of subjects or interfere with the conduct, progress, or completion of the study.
21. Abnormal thyroid function test during screening.
22. Screening or baseline cardiac troponin>ULN.

MAD

1. Special dietary requirements that cannot follow a unified diet.
2. Pregnant or lactating women who have a pregnancy plan during or within 3 months after the trial, female subjects tested positive for pregnancy during screening or baseline period.
3. Individuals with a history of febrile diseases or active infections within 7 days prior to the first administration of medication.
4. Positive urine drug screening results during screening or baseline period.
5. History of drug/drug abuse within 5 years prior to the start of the trial, or positive drug screening results during screening or baseline period.
6. Subjects who are receiving lipid-lowering treatment or have LDL-C>190 mg/dL and have a family history of coronary heart disease, arrhythmia, unexplained syncope, or cardiac arrest.
7. Existing history of QTc extension in the past:

   1. Screening period QTcF ≥ 450 ms.
   2. Family history of hypocalcemia or long QT interval syndrome.
   3. Using drugs that cause QT/QTc prolongation.
   4. Abnormal results of ECG with clinical significance determined by researchers.
8. Abnormal liver function: AST, ALT, ALP, GGT and TBIL>ULN.
9. Screening for smoking or using nicotine products within the first 3 months and during the study period.
10. Use of other investigational drugs 40 days prior to enrolment or within at least 5 half-lives of drug use.
11. Positive screening results for infectious diseases during the screening period, include HIV, HBsAg, HBcAb, HCV antibody Tests.
12. Any abnormal results of laboratory tests judged by the investigator to be clinically significant during the screening period.
13. Blood loss within 40 days prior to administration 50~500 mL, or loss of more than 500 mL of blood within 56 days prior to administration.
14. Men and women who consumed more than 1 unit per day prior to screening. [1 unit = 150 ml of wine, 360 ml of beer or 45 ml of 40% alcohol]. Subjects will not be permitted to consume alcohol 48 hours prior to dosing and while in the CRU.
15. Prescription and over-the-counter use within 14 days or at least 5 half-lives prior to the baseline period, or use of any drug or other substance that may affect CYP3A activity within 14 days or at least 5 half-lives before taking this study drug.
16. History of thyroid disease or clinically significant thyroid test abnormalities.
17. Allergy to thyroid medication.
18. Presence of any disease that may interfere with the absorption, distribution, metabolism or excretion of drugs, Including bile salt metabolism in the colon, such as gastrectomy, inflammatory bowel disease, etc.
19. According to the researcher's judgment, there are clinically significant diseases found, including but not limited to (gastrointestinal, kidney, liver, nervous, blood, endocrine, tumor, lung, immune, mental or cardiovascular diseases), researchers believe that participating in the study poses risks to participants.
20. Allergy to the investigational drug or any component of the investigational drug, Allergy history and constitution.
21. Diseases or conditions with clinical significance that researchers believe may pose a risk to the safety of subjects or interfere with the conduct, progress, or completion of the study.
22. Abnormal thyroid function test during screening.
23. Screening or baseline cardiac troponin>ULN.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-18 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Day1 to Day 28
  Physical examination, vital signs, including blood pressure, pulse, respiratory rate, and body temperature, 12 lead electrocardiogram, electrocardiogram monitoring, laboratory tests (including blood biochemistry, blood routine, urine routine, coagulation function).

SECONDARY OUTCOMES:
Single-Dose Pharmacokinetic (PK) Parameter (AUC0-∞) | Day 1
  Area under the concentration-time curve from time zero (pre-dose) extrapolation to infinite time.
Single-Dose Pharmacokinetic (PK) Parameter (AUC0-last) | Day 1
  AUC from time zero (pre-dose) to the time of the last measured concentration.
Single-Dose Pharmacokinetic (PK) Parameter (Cmax) | Day 1
  Maximum observed plasma concentration.
Single-Dose Pharmacokinetic (PK) Parameter (Tmax) | Day 1
  Time to the maximum plasma concentration.
Single-Dose Pharmacokinetic (PK) Parameter (T1/2) | Day 1
  Elimination half-life.
Single-Dose Pharmacokinetic (PK) Parameter (CL/F) | Day 1
  Apparent total plasma clearance.
Single-Dose Pharmacokinetic (PK) Parameter (Kel) | Day 1
  Elimination rate constant.
Single-Dose Pharmacokinetic (PK) Parameter (MRT) | Day 1
  Mean residence time.
Single-Dose Pharmacokinetic (PK) Parameter (Vz/F) | Day 1
  Apparent volume of distribution.
Multiple-Dose Pharmacokinetic (PK) Parameter (Ct_max) | Day 1, day 2, day 7, day 8, day 9, day 10, day 11, day 12, day 13, day 14, day 15.
  Maximum concentration during a dosing interva.
Multiple-Dose Pharmacokinetic (PK) Parameter (Ct_min) | Day 1, day 2, day 7, day 8, day 9, day 10, day 11, day 12, day 13, day 14, day 15.
  Minimum concentration during a dosing interval.
Multiple-Dose Pharmacokinetic (PK) Parameter (AUCtau) | Day 1, day 2, day 7, day 8, day 9, day 10, day 11, day 12, day 13, day 14, day 15.
  AUC over one dosing interval.
Multiple-Dose Pharmacokinetic (PK) Parameter (Tmax) | Day 1, day 2, day 7, day 8, day 9, day 10, day 11, day 12, day 13, day 14, day 15.
  Time to the maximum plasma concentration.
Multiple-Dose Pharmacokinetic (PK) Parameter (T1/2) | Day 1, day 2, day 7, day 8, day 9, day 10, day 11, day 12, day 13, day 14, day 15.
  Elimination half-life.
Multiple-Dose Pharmacokinetic (PK) Parameter (CL/F) | Day 1, day 2, day 7, day 8, day 9, day 10, day 11, day 12, day 13, day 14, day 15.
  Apparent total plasma clearance.
Multiple-Dose Pharmacokinetic (PK) Parameter (DF) | Day 1, day 2, day 7, day 8, day 9, day 10, day 11, day 12, day 13, day 14, day 15.
  Degree of fluctuation.
Multiple-Dose Pharmacokinetic (PK) Parameter (Ct_av) | Day 1, day 2, day 7, day 8, day 9, day 10, day 11, day 12, day 13, day 14, day 15.
  Mean plasma concentration during a dosing interval.
Multiple-Dose Pharmacokinetic (PK) Parameter (Rac) | Day 1, day 2, day 7, day 8, day 9, day 10, day 11, day 12, day 13, day 14, day 15.
  Accumulation factor.

OTHER OUTCOMES:
Pharmacodynamic (PD) Characteristics (Fasting serum LDL-C) | Day 1, day3, day 5, day 7, day 14, day 15, day 17.
  PD Characteristics of Multiple Oral Doses of CS060304 in Subjects with Elevated LDL-C
Pharmacodynamic (PD) Characteristics (HDL-C) | Day 1, day3, day 5, day 7, day 14, day 15, day 17.
  High-density lipoprotein cholesterol.
Pharmacodynamic (PD) Characteristics (TG) | Day 1, day 3, day 7, day 10, day 14, day 15, day 17.
  Triglyceride.
Pharmacodynamic (PD) Characteristics (TC) | Day 1, day3, day 5, day 7, day 14, day 15, day 17.
  Total cholesterol.
Pharmacodynamic (PD) Characteristics (Apo B) | Day 1, day3, day 5, day 7, day 14, day 15, day 17.
  Apolipoprotein B.
Pharmacodynamic (PD) Characteristics (SHBG) | Day 1, day3, day 7, day 10, day 14, day 15, day 17.
  Sex hormone binding globulin.
Thyroid function indicators (total serum T3) | Day 1, day3, day 7, day 10, day 14, day 15, day 17.
  Total serum T3.
Thyroid function indicators (T3) | Day 1, day3, day 7, day 10, day 14, day 15, day 17.
  Disassociate T3.
Thyroid function indicators (T4) | Day 1, day3, day 7, day 10, day 14, day 15, day 17.
  Thyroxine T4.
Thyroid function indicators (disassociate T4) | Day 1, day3, day 7, day 10, day 14, day 15, day 17.
  Disassociate T4.
Thyroid function indicators (TSH) | Day 1, day3, day 7, day 10, day 14, day 15, day 17.
  Thyroid stimulating hormone.
Drug concentration (QTcF) | Day 1, day 2.
  Orrected QT interval by Fridericia formula.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China